CLINICAL TRIAL: NCT07297667
Title: A Phase I Study of GCAR1, a Chimeric Antigen Receptor (CAR) T-CELL Therapy for Participants With Selected Relapsed/Refractory GPNMB-Expressing Solid Tumours
Brief Title: GCAR1, a Chimeric Antigen Receptor (CAR) T-CELL Therapy for Relapsed/Refractory GPNMB-Expressing Solid Tumours
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Canadian Cancer Trials Group (Network)
Collaborators: University of Calgary (Other); Canadian Institutes of Health Research (CIHR) (Other Government); BioCanRx (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I246
Record Dates: First submitted 2025-12-09; First posted 2025-12-22 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Alveolar Soft Part Sarcoma; Renal Cell Carcinoma; Triple Negative Breast Cancer
MeSH Terms: conditions — Sarcoma, Alveolar Soft Part; Carcinoma, Renal Cell; Triple Negative Breast Neoplasms | interventions — fludarabine; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GCAR1 Infusion (Experimental)
  Interventions: Drug: Fludarabine; Drug: Cyclophosphamide; Biological: GCAR1

INTERVENTIONS:
Drug: Fludarabine — Assigned at enrollment
Drug: Cyclophosphamide — Assigned at enrollment
Biological: GCAR1 — Dose escalation

SUMMARY:
The purpose of this study is to identify the highest dose of GCAR1, a chimeric antigen receptor (CAR-T) cell therapy, that can be tolerated without causing very severe side effects, and to see what effects GCAR1 has on selected cancers

DETAILED DESCRIPTION:
GCAR1 is a type of CAR-T cell therapy that is designed to identify a protein (GPNMB) that is present on the cells of certain types of cancer. Laboratory tests have shown that GCAR1 helps the immune system recognize cancer cells and may help slow down cancer growth.

The purpose of this study is to find out what effects the new treatment, GCAR1 has on certain cancers. This study will test increasing doses of GCAR1 in participants with alveolar soft part sarcoma (ASPS), triple negative breast cancer (TNBC), and renal cell carcinoma (RCC) expressing high levels of the GPNMB protein, to establish recommended doses for further testing.

ELIGIBILITY:
Inclusion Criteria:

* Archival tumour specimen must be positive for GPNMB with high expression by immunohistochemistry (central laboratory testing).
* Histologically and/or cytologically confirmed diagnosis of one of the following tumours that is advanced/ metastatic/ recurrent or unresectable, for which no curative therapy exists.
* alveolar soft part sarcoma
* renal cell carcinoma (excluding clear cell)
* triple negative breast cancer (ER, PR and HER-2 negative as defined by ASCO/CAP criteria)
* Must have a formalin fixed paraffin embedded tissue block (from primary or metastatic tumour) available and must have provided informed consent for the release of the block.
* Presence of radiologically documented disease.
* Measurable disease as defined by RECIST 1.1.
* ASPS participants ≥ 15 years of age.
* TNBC and RCC participants ≥ 18 years of age.
* ECOG performance status of 0 or 1 or Karnofsky or Lansky > 60.
* Anticipated life expectancy of ≥ 6 months.
* Must have received prior systemic therapy as shown below;
* ASPS - completed all systemic therapy available that has been shown to improve survival (unless contraindicated).
* TNBC

  1. Progressive disease following at least one line of systemic treatment for metastatic disease which must include an ADC (all participants) and an ICI (participants whose tumours express PD-L1).
  2. ≤3 lines of treatment for metastatic disease.
  3. Must have had at least 1 prior line of cytotoxic chemotherapy for breast cancer, in any setting, which must have included an anthracycline and a taxane (unless contraindicated).
* RCC - must have progressive disease following at least one line of systemic treatment for metastatic disease that must have included an ICI and a VEGFR targeted agent (unless contraindicated).
* Participants must have recovered to ≤ grade 1 from all reversible toxicity related to prior therapies.
* Adequate washout must be followed per protocol.
* Previous major surgery is permitted ≥21 days prior to enrollment
* Prior external beam radiation is permitted ≥28 prior to enrollment. Concurrent radiotherapy is not permitted.
* Adequate hematologic and biochemical parameters.
* Consent and assent, when applicable, must be appropriately obtained in accordance with applicable local and regulatory requirements. Each participant or their parent/ legal guardian (if applicable) must sign a consent form prior to screening onto the trial to document their willingness to participate.
* Fit for leukapheresis and has adequate venous access for cell collection.
* Must be accessible for treatment and follow up at the participating centre for a minimum of 12 months or for as long as is deemed necessary by the treating physician.
* Participants of childbearing potential must have agreed to use a highly effective contraceptive method.

Exclusion criteria

* Participants on active anticancer therapy for other advanced or metastatic malignancies.
* Concurrent treatment with other anti-cancer therapy
* Prior therapy with a gene therapy product or any adoptive T cell therapy or prior GPNMB targeting therapy.
* Live attenuated vaccination administered within 30 days prior to or planned within 30 days after GCAR1 therapy.
* Primary immunodeficiency or history of severe autoimmune disease (including: Crohn's disease, rheumatoid arthritis, systemic lupus) requiring immunosuppressive agents/ systemic disease modifying agents within 2 years of enrollment.
* Active or uncontrolled infections or with serious illnesses or medical conditions which would not permit the participant to be managed according to the protocol including but not limited to:
* Hepatitis B or C virus (HBV or HCV). For participants with previous HBV or HCV infection who are currently on treatment, they are eligible if they have an undetectable viral load via quantitative PCR and/or nucleic acid testing
* HIV positive by serology and PCR
* Uncontrolled fungal, bacterial, viral or other infection
* Current infection with HTLV-1
* Tuberculosis
* Syphilis
* West Nile Virus
* Untreated and/or uncontrolled cardiovascular conditions and/or symptomatic cardiac dysfunction (including cardiac ventricular arrhythmias requiring medication, history of 2nd or 3rd degree atrioventricular conduction defects) or unstable angina congestive heart failure or myocardial infarction within the previous year.
* Known sensitivity or allergy to fludarabine, cyclophosphamide or any of their components, or to GCAR1 or any of its components.
* Active intracerebral metastases or leptomeningeal disease. Participants who have received definitive treatment, are clinically stable and do not require corticosteroids are eligible to participate in the trial.
* Pregnant or breastfeeding women.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2028-12-01 (Estimated); Study Completion 2033-09-01 (Estimated)

PRIMARY OUTCOMES:
To determine the recommended phase II dose (RP2D), defined as the next lower dose below the maximum administered dose, of GPNMB directed CAR T cell therapy | 3 years
  (GCAR1) in participants with selected tumours (alveolar soft part sarcoma, renal cell carcinoma (excluding clear cell), triple negative breast cancer) expressing GPNMB

SECONDARY OUTCOMES:
Number and severity of adverse eventsGCAR1 utilizing CTCAE v5.0 | 3 years
Overall response rate utilizing RECIST 1.1 | 3 years
Duration of response | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Mona Shafey, Study Chair — Tom Baker Cancer Centre, Calgary, Alberta, Canada
Locations (3):
- Canada (3):
  - Arthur J.E. Child Comprehensive Cancer Centre, Calgary, Alberta
  - Ottawa Hospital Research Institute, Ottawa, Ontario
  - University Health Network Princess Margaret Hospital, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: Yes
According to CCTG Policies
URL: https://www.ctg.queensu.ca/public/policies